CLINICAL TRIAL: NCT00235833
Title: Long-term Continuously Repeated Dose Study of Adalimumab (D2E7) in Patients With Rheumatoid Arthritis
Brief Title: Adalimumab in Adult Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry); Eisai Co., Ltd. (Industry)
Responsible Party: Eiichi Makino, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-564
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 40 mg eow (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg every other week (eow), subcutaneous (sc)
  Other Names: ABT-D2E7; Humira

SUMMARY:
The purpose of the study is to assess the long-term safety, tolerability, and efficacy of repeated administration of adalimumab in adult Japanese subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the prior adalimumab study
* Body weight less than 100 kg.
* Subject's who wished to continue the study drug administration
* Females must be postmenopausal for at least 1 year, surgically sterile, or practicing birth control throughout the study and for 90 days after study completion.

Exclusion Criteria:

* A subject who experienced any of the following during the prior adalimumab sc dosing study:

  * Advanced or poorly controlled diabetes
  * Any poorly controlled medical condition
  * Intra-articular, intramuscular or iv administration of corticosteroids
  * Joint surgery.
* A subject who has been prescribed excluded medications during previous adalimumab study.
* History of clinically significant drug or alcohol abuse, intravenous (iv) drug abuse, active infection with listeria or tuberculosis (TB), lymphoma, leukemia, or any malignancy with the exception of successfully treated non- metastatic basal cell carcinoma of the skin.
* A subject who experienced chronic or active infection or any major episode of infection requiring hospitalization or treatment with intravenous (iv) antibiotics within 30 days of entry into study or chronic use of oral antibiotics within 14 days of entry into study.
* Preexisting or recent onset of central nervous system (CNS) demyelinating disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-06; Primary Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Hashimoto, Ph.D., Study Director — Abbott
Locations (7):
- Japan (7):
  - Tokyo, Metropolis
  - Fukuoka, Prefecture
  - Hiroshima, Prefecture
  - Ibaraki, Prefecture
  - Nagasaki, Prefecture
  - Osaka, Prefecture
  - Saitama, Prefecture

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese subjects with moderate to severe rheumatoid arthritis (RA) in relatively good physical health excluding RA symptoms and who completed a preceding continuous repeated administration study of adalimumab (DE035X/D2E7-J081-003) who wished to continue treatment until approval of adalimumab in Japan.
Groups:
- Adalimumab 40 mg Eow: Adalimumab 40 mg subcutaneously (sc) administered every other week (eow) until approval of adalimumab in Japan.
Period: Overall Study
Arm/Group | Adalimumab 40 mg Eow
Started | 25
Completed | 9
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4
Region of Enrollment [Number; unit: participants]
  Japan | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders With American College of Rheumatology (ACR) Criteria Improvement of at Least 20%, 50%, and 70% (ACR 20/50/70 Responders)
Description: Number of subjects with American College of Rheumatology (ACR) criteria improvement consisting of 20%, 50%, and 70% (ACR20, ACR50, and ACR70, respectively) reduction in tender or swollen joint counts [TJC or SJC, respectively] and 20%, 50%, and 70% improvement, respectively, in 3 of the following 5 criteria: [1] physician's global assessment of disease activity [PGA], [2] subject's assessment of disease activity, [3] subject's assessment of pain, [4] subject's assessment of functional disability via a health assessment questionnaire [HAQ], and [5] C-reactive protein [CRP]) at each visit
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Population: Analysis was based on observed data.
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
participants
  Week 0 ACR20 | 12
  Week 0 ACR50 | 7
  Week 0 ACR70 | 5
  Week 6 ACR20 | 15
  Week 6 ACR50 | 12
  Week 6 ACR70 | 5
  Week 12 ACR20 | 16
  Week 12 ACR50 | 11
  Week 12 ACR70 | 6
  Week 18 ACR20 | 18
  Week 18 ACR50 | 11
  Week 18 ACR70 | 7
  Week 24 ACR20 | 16
  Week 24 ACR50 | 11
  Week 24 ACR70 | 4
  Week 36 ACR20 | 15
  Week 36 ACR50 | 10
  Week 36 ACR70 | 6
  Week 48 ACR20 | 13
  Week 48 ACR50 | 10
  Week 48 ACR70 | 5
  Week 60 ACR20 | 12
  Week 60 ACR50 | 11
  Week 60 ACR70 | 6
  Week 72 ACR20 | 11
  Week 72 ACR50 | 10
  Week 72 ACR70 | 3
  Week 84 ACR20 | 11
  Week 84 ACR50 | 9
  Week 84 ACR70 | 7
  Week 96 ACR20 | 11
  Week 96 ACR50 | 10
  Week 96 ACR70 | 6
  Week 108 ACR20 | 11
  Week 108 ACR50 | 10
  Week 108 ACR70 | 6
  Week 120 ACR20 | 10
  Week 120 ACR50 | 10
  Week 120 ACR70 | 6
  Week 132 ACR20 | 10
  Week 132 ACR50 | 7
  Week 132 ACR70 | 5
  Week 144 ACR20 | 10
  Week 144 ACR50 | 9
  Week 144 ACR70 | 7
  Week 156 ACR20 | 9
  Week 156 ACR50 | 8
  Week 156 ACR70 | 4
  Week 168 ACR20 | 9
  Week 168 ACR50 | 8
  Week 168 ACR70 | 6
  Week 180 ACR20 | 10
  Week 180 ACR50 | 9
  Week 180 ACR70 | 5
  Week 192 ACR20 | 9
  Week 192 ACR50 | 8
  Week 192 ACR70 | 5
  Week 204 ACR20 | 10
  Week 204 ACR50 | 8
  Week 204 ACR70 | 4
  Week 216 ACR20 | 9
  Week 216 ACR50 | 8
  Week 216 ACR70 | 4
  Week 228 ACR20 | 9
  Week 228 ACR50 | 7
  Week 228 ACR70 | 3
  Week 240 ACR20 | 7
  Week 240 ACR50 | 4
  Week 240 ACR70 | 1
  Week 252 ACR20 | 5
  Week 252 ACR50 | 3
  Week 252 ACR70 | 2
  Week 264 ACR20 | 2
  Week 264 ACR50 | 1
  Week 264 ACR70 | 1
  Final Value ACR20 | 13
  Final Value ACR50 | 11
  Final Value ACR70 | 8

2. Secondary Outcome: Mean Change From Baseline in Tender Joint Count (TJC, Max = 68), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (last assessment in preceding study prior to adalimumab injection) in tender joint count (TJC, max = 68), a component of the ACR criteria, by visit
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: TJC
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
TJC
  Week 0 | -11.2 (14.5)
  Week 6 | -13.4 (11.2)
  Week 12 | -16.0 (14.0)
  Week 18 | -17.5 (12.2)
  Week 24 | -16.3 (13.7)
  Week 36 | -17.0 (13.4)
  Week 48 | -18.1 (13.8)
  Week 60 | -18.5 (13.2)
  Week 72 | -18.1 (13.2)
  Week 84 | -21.9 (13.7)
  Week 96 | -22.8 (13.6)
  Week 108 | -21.8 (13.6)
  Week 120 | -22.7 (14.4)
  Week 132 | -22.0 (14.5)
  Week 144 | -21.2 (14.4)
  Week 156 | -22.1 (14.9)
  Week 168 | -22.7 (13.6)
  Week 180 | -22.7 (13.5)
  Week 192 | -23.3 (14.5)
  Week 204 | -23.1 (14.7)
  Week 216 | -23.7 (14.7)
  Week 228 | -23.4 (14.7)
  Week 240 | -24.6 (13.7)
  Week 252 | -26.7 (17.5)
  Week 264 | -25.0 (7.1)
  Final Value | -15.8 (13.8)

3. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count (SJC, Max = 66), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline(last assessment in preceding study prior to adalimumab injection) in the SJC (max = 66) component of the ACR criteria
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: SJC
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
SJC
  Week 0 | -8.8 (11.0)
  Week 6 | -11.3 (11.3)
  Week 12 | -12.0 (12.1)
  Week 18 | -14.4 (9.6)
  Week 24 | -13.8 (10.7)
  Week 36 | -12.4 (6.8)
  Week 48 | -14.9 (6.3)
  Week 60 | -14.8 (5.7)
  Week 72 | -14.5 (6.5)
  Week 84 | -13.5 (4.7)
  Week 96 | -13.9 (5.8)
  Week 108 | -13.8 (5.7)
  Week 120 | -13.2 (4.5)
  Week 132 | -13.2 (4.2)
  Week 144 | -14.0 (3.9)
  Week 156 | -13.3 (4.3)
  Week 168 | -13.2 (5.5)
  Week 180 | -13.7 (4.4)
  Week 192 | -13.4 (4.9)
  Week 204 | -12.9 (5.3)
  Week 216 | -12.6 (5.8)
  Week 228 | -12.9 (5.5)
  Week 240 | -11.8 (5.8)
  Week 252 | -11.8 (5.8)
  Week 264 | -12.0 (8.5)
  Final Value | -10.1 (11.8)

4. Secondary Outcome: Mean Change From Baseline in Physician's Global Assessment of Disease Activity (PGA) Using a Visual Analog Scale (0 - 100 mm With 100 mm Being the Worst Possible Assessment), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (last assessment in preceding study prior to adalimumab injection) in PGA (a visual analog scale from 0 - 100 mm with 100 mm being the worst possible assessment), a component of the ACR criteria, by visit.
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: mm on scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
mm on scale
  Week 0 | -27.0 (28.6)
  Week 6 | -34.5 (28.4)
  Week 12 | -40.7 (22.0)
  Week 18 | -42.2 (22.1)
  Week 24 | -41.3 (24.2)
  Week 36 | -34.3 (19.9)
  Week 48 | -40.7 (21.7)
  Week 60 | -39.2 (27.8)
  Week 72 | -39.2 (26.7)
  Week 84 | -40.1 (29.8)
  Week 96 | -51.7 (20.9)
  Week 108 | -50.6 (20.6)
  Week 120 | -50.5 (27.3)
  Week 132 | -50.1 (21.1)
  Week 144 | -43.6 (28.1)
  Week 156 | -47.2 (28.9)
  Week 168 | -49.5 (25.6)
  Week 180 | -51.8 (24.4)
  Week 192 | -49.6 (26.7)
  Week 204 | -47.5 (22.7)
  Week 216 | -52.5 (22.8)
  Week 228 | -49.5 (23.2)
  Week 240 | -47.3 (18.9)
  Week 252 | -51.7 (23.5)
  Week 264 | -35.5 (38.9)
  Final Value | -31.2 (32.7)

5. Secondary Outcome: Mean Change From Baseline in Subject's Global Assessment of Disease Activity Using a Visual Analog Scale (0 - 100 mm With 100 mm Being the Worst Possible Assessment), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (last assessment in preceding study prior to adalimumab injection) in subject's global assessment of disease activity (a visual analog scale from 0 - 100 mm with 100 mm being the worst case), a component of the ACR criteria, by visit
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: mm on scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
mm on scale
  Week 0 | -21.7 (27.4)
  Week 6 | -29.5 (25.8)
  Week 12 | -33.3 (25.8)
  Week 18 | -35.1 (25.7)
  Week 24 | -35.6 (22.2)
  Week 36 | -33.0 (24.5)
  Week 48 | -38.3 (24.3)
  Week 60 | -38.7 (26.4)
  Week 72 | -39.3 (24.9)
  Week 84 | -37.1 (30.3)
  Week 96 | -42.9 (26.0)
  Week 108 | -35.1 (31.0)
  Week 120 | -40.4 (26.2)
  Week 132 | -34.1 (21.3)
  Week 144 | -37.3 (26.4)
  Week 156 | -34.5 (31.1)
  Week 168 | -37.2 (26.3)
  Week 180 | -36.1 (20.4)
  Week 192 | -35.3 (26.1)
  Week 204 | -35.0 (18.0)
  Week 216 | -30.3 (23.9)
  Week 228 | -30.7 (27.6)
  Week 240 | -23.9 (22.4)
  Week 252 | -25.0 (21.2)
  Week 264 | -19.5 (10.6)
  Final Value | -20.0 (27.9)

6. Secondary Outcome: Mean Change From Baseline (Last Assessment in Preceding Study Prior to Adalimumab Injection) in Subject's Assessment of Pain Using a Visual Analog Scale (0 - 100 mm With 100 mm Being the Worst Possible Pain), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (last assessment in preceding study prior to adalimumab injection) in subject's assessment of pain (using a visual analog scale from 0 - 100 mm with 100 mm being the worst possible pain), a component of the ACR criteria, by visit
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: mm on scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
mm on scale
  Week 0 | -13.7 (31.6)
  Week 6 | -23.1 (24.7)
  Week 12 | -27.2 (27.3)
  Week 18 | -29.1 (28.2)
  Week 24 | -30.6 (20.2)
  Week 36 | -26.2 (28.2)
  Week 48 | -32.7 (22.2)
  Week 60 | -33.4 (26.1)
  Week 72 | -33.4 (24.2)
  Week 84 | -32.9 (26.7)
  Week 96 | -37.6 (22.7)
  Week 108 | -31.8 (27.6)
  Week 120 | -35.0 (21.9)
  Week 132 | -30.0 (18.6)
  Week 144 | -33.1 (24.1)
  Week 156 | -29.9 (31.0)
  Week 168 | -31.8 (24.0)
  Week 180 | -32.8 (19.8)
  Week 192 | -31.0 (23.4)
  Week 204 | -30.6 (17.4)
  Week 216 | -24.4 (23.7)
  Week 228 | -26.5 (26.8)
  Week 240 | -24.9 (23.7)
  Week 252 | -20.3 (24.4)
  Week 264 | -7.0 (2.8)
  Final Value | -14.4 (29.6)

7. Secondary Outcome: Mean Change From Baseline in Disability Index of the Health Assessment Questionnaire [HAQ], a Component the of ACR Criteria, by Visit
Description: Mean change from baseline (last assessment in preceding study prior to adalimumab injection) in disability index of the health assessment questionnaire [HAQ; includes 20 questions assessing physical function in 8 domains. The questions are evaluated on a scale from 0 - 3 to measure the ability to perform certain activities (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do so).], a component the of ACR criteria, by visit
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
units on a scale
  Week 0 | -0.41 (0.77)
  Week 6 | -0.48 (0.64)
  Week 12 | -0.47 (0.65)
  Week 18 | -0.50 (0.72)
  Week 24 | -0.49 (0.76)
  Week 36 | -0.43 (0.77)
  Week 48 | -0.63 (0.72)
  Week 60 | -0.66 (0.81)
  Week 72 | -0.73 (0.81)
  Week 84 | -0.82 (0.71)
  Week 96 | -0.80 (0.71)
  Week 108 | -0.74 (0.83)
  Week 120 | -0.73 (0.81)
  Week 132 | -0.63 (0.80)
  Week 144 | -0.63 (0.80)
  Week 156 | -0.58 (0.69)
  Week 168 | -0.64 (0.78)
  Week 180 | -0.63 (0.70)
  Week 192 | -0.49 (0.73)
  Week 204 | -0.51 (0.67)
  Week 216 | -0.51 (0.77)
  Week 228 | -0.49 (0.93)
  Week 240 | -0.36 (0.70)
  Week 252 | -0.25 (0.80)
  Week 264 | 0.25 (1.41)
  Final Value | -0.31 (0.77)

8. Secondary Outcome: Mean Change From Baseline in C-reactive Protein [CRP; mg/dL], a Component of the ACR Criteria, by Visit.
Description: Mean change from baseline (last assessment in preceding study prior to adalimumab injection) in C-reactive protein [CRP; mg/dL], a component of the ACR criteria, by visit.
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
mg/dL
  Week 0 | -0.92 (2.64)
  Week 6 | -2.30 (2.73)
  Week 12 | -2.49 (3.55)
  Week 18 | -2.11 (3.22)
  Week 24 | -2.62 (2.49)
  Week 36 | -2.42 (3.17)
  Week 48 | -2.94 (3.37)
  Week 60 | -3.31 (3.15)
  Week 72 | -3.05 (3.35)
  Week 84 | -2.84 (3.50)
  Week 96 | -3.37 (3.08)
  Week 108 | -3.07 (3.09)
  Week 120 | -3.16 (3.62)
  Week 132 | -3.23 (3.39)
  Week 144 | -3.14 (3.66)
  Week 156 | 0.01 (10.96)
  Week 168 | -3.47 (3.42)
  Week 180 | -3.49 (3.28)
  Week 192 | -3.21 (3.42)
  Week 204 | -3.30 (3.22)
  Week 216 | -2.90 (2.57)
  Week 228 | -2.93 (2.57)
  Week 240 | -1.71 (6.10)
  Week 252 | -1.89 (3.56)
  Week 264 | -4.16 (5.35)
  Final Value | -1.14 (4.23)

9. Secondary Outcome: Area Under the Curve (AUC; From Start of the Study to Each Study Visit) of Subjects' Who Improved at Least 20% in ACR Response Criteria (ACR20 Response)
Description: Sum of the duration (from start of study to each study visit) when a subject with American College of Rheumatology (ACR) criteria improved by 20% (ACR20) in tender or swollen joint counts [TJC or SJC, respectively] and 20% improvement in 3 of the following 5 criteria: [1] Physician's global assessment (PGA), [2] subject's assessment of disease activity, [3] subject's assessment of pain, [4] subject's assessment of functional disability via a health assessment questionnaire [HAQ], and [5] C-reactive protein (CRP)
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 25
Weeks
  Week 0 - Week 6 | 3.2 (2.7)
  Week 0 - Week 12 | 7.0 (5.5)
  Week 0 - Week 18 | 11.0 (8.0)
  Week 0 - Week 24 | 15.1 (10.6)
  Week 0 - Week 36 | 22.6 (15.9)
  Week 0 - Week 48 | 29.3 (21.1)
  Week 0 - Week 60 | 35.3 (26.3)
  Week 0 - Week 72 | 40.8 (31.3)
  Week 0 - Week 84 | 46.1 (36.2)
  Week 0 - Week 96 | 51.4 (41.3)
  Week 0 - Week 108 | 56.6 (46.7)
  Week 0 - Week 120 | 61.7 (52.0)
  Week 0 - Week 132 | 66.5 (57.2)
  Week 0 - Week 144 | 71.3 (62.5)
  Week 0 - Week 156 | 75.8 (67.7)
  Week 0 - Week 168 | 80.2 (72.7)
  Week 0 - Week 180 | 84.7 (78.0)
  Week 0 - Week 192 | 89.3 (83.4)
  Week 0 - Week 204 | 93.8 (88.2)
  Week 0 - Week 216 | 98.4 (92.7)
  Week 0 - Week 228 | 102.7 (97.1)
  Week 0 - Week 240 | 106.6 (101.0)
  Week 0 - Week 252 | 109.4 (104.2)
  Week 0 - Week 264 | 111.1 (106.4)

10. Secondary Outcome: Number of Subjects With Morning Stiffness at Each Visit
Description: The number of subjects with morning stiffness (assessed as present or absent) at each visit among those who had morning stiffness at baseline (21).
Time Frame: Every 6 weeks up to Week 24 and every 12 weeks thereafter up to study completion or discontinuation (final value)
Population: Subjects analyzed (as-observed) include only those who had morning stiffness at baseline.
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 21
participants
  Week 0 | 16
  Week 6 | 15
  Week 12 | 11
  Week 18 | 11
  Week 24 | 9
  Week 36 | 10
  Week 48 | 6
  Week 60 | 5
  Week 72 | 7
  Week 84 | 6
  Week 96 | 4
  Week 108 | 4
  Week 120 | 3
  Week 132 | 3
  Week 144 | 3
  Week 156 | 3
  Week 168 | 2
  Week 180 | 2
  Week 192 | 3
  Week 204 | 4
  Week 216 | 3
  Week 228 | 3
  Week 240 | 3
  Week 252 | 2
  Week 264 | 1
  Final Value | 15

ADVERSE EVENTS:
Arm/Group | Adalimumab 40 mg Eow
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Eow (N=25)
Lymphadenitis (Blood and lymphatic system disorders) | 1
Brugada syndrome (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Eow (N=25)
Diarrhoea (Gastrointestinal disorders) | 6
Dental caries (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Enterocolitis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 2
Adverse drug reaction (General disorders) | 4
Chest pain (General disorders) | 2
Injection site reaction (General disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 4
Nasopharyngitis (Infections and infestations) | 15
Cystitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tinea blanca (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Arthropod sting (Injury, poisoning and procedural complications) | 3
Animal bite (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 2
Blood glucose increased (Investigations) | 3
DNA antibody positive (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 2
Lymphocyte percentage decreased (Investigations) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 3
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Due to the small population, statistical tests were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; most restrictive agreement states Medical Institution shall not disclose materials/information disclosed by Abbott Japan in connection with the Clinical Research, or information obtained by conducting the Clinical Research, to third parties without Abbott Japan's prior written approval. When Medical Institution intends to publish information obtained by conducting the Clinical Research, Medical Institution shall obtain Abbott Japan's prior written approval.